CLINICAL TRIAL: NCT06435988
Title: The Effect of the Training Given Using the Pecha Kucha Technique on the Anxiety and Birth Satisfaction of the First Pregnant Women Followed in Labor.
Brief Title: The Effect of Training With Pecha Kucha on Anxiety and Birth Satisfaction in Pregnant Women.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hatice Gamze Recber, principal ınvestigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HGRecber
Record Dates: First submitted 2024-05-14; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: First Pregnancy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no ıntervention (No Intervention): no ıntervention
- experimental (Experimental): Training in the pecha kucha technique
  Interventions: Behavioral: Training in the pecha kucha technique

INTERVENTIONS:
Behavioral: Training in the pecha kucha technique — Providing labor training to pregnant women with the Pecha Kucha technique
  Arms: experimental

SUMMARY:
For this purpose, the distribution of Pecha Kucha user's birth information education on state/trait anxiety and birth hope in primiparous pregnant women is determined.

The main question the researcher aims to answer is:

Do anxiety and birth changes in pregnant women who receive Pecha Kucha's registered birth information training? There are 25 pregnant women in the experimental and 25 control groups. After the training, participants in the experimental groups will answer the satisfaction survey and questions about trait anxiety.

DETAILED DESCRIPTION:
The research was started after receiving ethics committee approval and written approval from the relevant institution. Pechka kucha presentation was prepared by the researcher in accordance with the literature information and the features required by the technique. For the content validity of the travay information presentation prepared with the PK technique, expert opinions were received from 10 academicians who have scientific studies on this subject.

After receiving expert approval of the presentation, the data collection process began. The research population consists of primiparous pregnant women who were admitted to the delivery room and followed during birth. The participants included in the study were assigned to groups through randomization, ensuring homogeneity in the distribution of the groups. "Random Allocation Software Program" was used to randomize the participants into groups, and the randomization list of the study was created by determining the number of each participant and the number of groups.

Participants admitted to the delivery room for normal birth, in the order on the randomization list; were assigned as a control and an experimental group by the researcher.

Only participants assigned to the randomization group were studied until completion. After the birth of the participants was completed, the first participant who was admitted to the delivery room and met the research criteria was assigned to the other group on the randomization list and the necessary interventions were carried out. If the participant has a cesarean section during the study or leaves the study for any reason; The first participant admitted to the delivery room and meeting the research criteria will be assigned to the other group on the randomization list.

The research was explained to the participant assigned to the experimental group, and if voluntary participation was required, the 'Informed Consent Form' was signed.

Participants in the experimental group were given 'Pecha Kucha Travay Information' training. The presentation was held in the TDL (Labor-Delivery-Postpartum) unit, in single rooms, with a seating arrangement facing each other. The presentation was made on the researcher's tablet with an 8-inch screen size. The position of the tablet was adjusted to the middle point in the seating arrangement of the participant and the researcher. Before the training, he was informed about the duration of the presentation and it was stated that he could talk about the questions he wanted to ask at the end of the presentation.

The presentation, prepared with the Pechka Kucha method and lasting 6 minutes and 20 seconds, was explained to the participant via tablet. Then, the introductory information form and the state-trait anxiety scale were filled out. After birth, participants in the experimental group filled out the 'Birth Satisfaction Scale' before being transferred from the delivery room to the ward.

ELIGIBILITY:
Inclusion Criteria:

* Primary pregnant women,
* Pregnant women aged 18 and over,
* Pregnant women in the latent phase of labor
* Pregnant women who do not have perinatological risk,
* Pregnant women who can understand and speak Turkish

Exclusion Criteria:

* • Risky pregnant women,

  * Pregnant woman in active phase,
  * Pregnant women who develop an obstetric complication during labor follow-up (Fetal distress, Cord prolapse, Uterine hyperstimulation, non-progressive labor, malpresentation, etc.).
  * There is a problem that prevents communication

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
State and Trait Anxiety ScaleWomen. | 24 hours
  After the total weights of the direct and reversed expressions are found separately, the total weight score of the reverse expressions is subtracted from the total weight score obtained for the direct expressions. A predetermined and unchanging value is added to this number. This constant value is 50 for the State Anxiety Scale and 35 for the Trait Anxiety Scale. The final value obtained represents the individual's anxiety score.
Birth Experience Scale | 24 hours
  The scale, which was developed to measure women's birth experience in different dimensions, has four sub-dimensions and 22 items. The first 19 items of the scale are evaluated using a four-point scale and the last three items are evaluated using VAS. In DSS, the first 19 items are scored from 1 to 4; I completely agree = 1, I mostly agree = 2, I partially agree = 3, I completely disagree = 4.
  The scores on the VAS scale are categorical; It is classified as 0-40 = 1, 41-60 = 2, 61-80 = 3, 81-100 = 4. Cronbach's alpha value of the scale; 0.56 for the Birth Process sub-dimension, 0.73 for the Professional Support/Help subscale, 0.63 for the Perceived Security/Memories subscale, 0.64 for Participation in Decisions sub-dimension The total scale Cronbach alpha reliability coefficient was found to be 0.76.

CONTACTS AND LOCATIONS:
Overall Officials: resmiye özdilek, Asst.Prof., Study Director — Kocaeli University Faculty of Health Sciences
Locations (1):
- Kocaeli Üniversitesi, Gebze, Kocaeli̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No